CLINICAL TRIAL: NCT01098656
Title: A Phase III Study of Lenalidomide Maintenance After Debulking Therapy in Patients With Advanced Cutaneous T-Cell Lymphoma
Brief Title: Lenalidomide Maintenance Post-debulking in Advanced CTCL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruitment prematurely halted following company's decision to stop financial support to the study
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-21081; EU-21020; 2009-011020-65 (EudraCT Number); CELGENE-EORTC-21081
Record Dates: First submitted 2010-04-02; First posted 2010-04-05 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Lymphoma
Keywords: stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Mycosis Fungoides; Sezary Syndrome; Lymphoma, T-Cell, Cutaneous | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lenalidomide (Experimental)
  Interventions: Drug: lenalidomide
- Observation (No Intervention)

INTERVENTIONS:
Drug: lenalidomide — The starting dose of lenalidomide is 25 mg orally once daily on days 1-21 of repeated 28-day cycles.
  Dosing is continued or modified based upon clinical and laboratory findings (dose reductions: 20 mg, 15 mg, 10 mg and 5 mg)
  Arms: lenalidomide

SUMMARY:
RATIONALE: Observation is watching a patient's condition but not giving treatment unless symptoms appear or change. Lenalidomide may stop the growth of cancer cells by blocking blood flow to the cancer. It is not yet known whether observation or lenalidomide is more effective in treating patients who are in complete or partial response after receiving previous gemcitabine hydrochloride or doxorubicin hydrochloride liposome for cutaneous T-cell lymphoma or mycosis fungoides/Sézary syndrome.

PURPOSE: This randomized phase III trial is studying observation to see how well it works compared with lenalidomide in treating patients who are in complete or partial response after receiving previous gemcitabine hydrochloride or doxorubicin hydrochloride liposome for stage IIB, stage III, or stage IV cutaneous T-cell lymphoma or stage IIB, stage III, or stage IV mycosis fungoides/Sézary syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if observation versus lenalidomide maintenance therapy after debulking with gemcitabine hydrochloride or pegylated liposomal doxorubicin hydrochloride with or without radiotherapy prolongs progression-free survival of patients with advanced stage IIIB or IV T-cell cutaneous lymphoma or mycosis fungoides/Sézary syndrome not previously treated with other intravenous chemotherapy.

OUTLINE: This is a multicenter study. Patients are stratified according to institution, response to debulking treatment (complete response vs partial response), and disease (mycosis fungoides [MF] vs erythrodermic MF/Sézary syndrome). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Beginning 4-6 weeks after completion of prior debulking therapy, patients undergo observation for 560 days.
* Arm II: Beginning 4-6 weeks after completion of prior debulking therapy, patients receive oral lenalidomide once a day on days 1-21. Treatment repeats every 28 days for 20 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 4 weeks and then every 12 weeks thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnoses of advanced T-cell cutaneous lymphoma or mycosis fungoides/Sézary syndrome

  * Stage IIB-IV disease
* Achieved complete or partial response after undergoing prior debulking therapy with 1 of the following recommended* regimens with or without radiotherapy**:

  * Gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 of a 28-day course at a dose of 1,000 to 1,200 mg/m² for a total of four courses
  * Pegylated liposomal doxorubicin hydrochloride IV over 1 hour on days 1 and 15 of a 28-day course at a dose of 20 mg/m² for a total of four courses NOTE: *These recommended regimens can be altered according to local institutional policies. In case of drug intolerance, the study regimen can be switched from one regimen to the other.

NOTE: **Local low-dose/energy-ionizing radiation therapy allowed as part of the debulking process to treat lesions that do not respond after 3 courses of debulking chemotherapy.

* Sézary cell burden must be decreased by at least 50% after debulking in patients with Sézary syndrome
* Disease not appropriate for skin-directed therapy per local institution standards
* No disease progression between registration and randomization
* No CNS involvement

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy > 12 months
* Hemoglobin ≥ 10 g/dL
* Absolute neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 60 x 10^9/L
* Total bilirubin ≤ 1.5 times upper limit of normal (UNL)
* Alkaline phosphatase ≤ 3 times UNL
* ALT/AST ≤ 3 times UNL
* Electrolytes (including sodium, potassium, and chloride) normal
* Creatinine normal
* Creatinine clearance ≥ 60 mL/min
* Uric acid and calcium normal
* Free T4 and TSH ≤ 1.5 times ULN
* Patients with a buffer range from the normal values of +/- 10% for hematology and biochemistry are acceptable
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception 4 weeks prior to, during, and for 4 weeks after completion of study therapy
* Males must agree not to donate semen during and for 1 week after completion of study therapy
* Patients with high risk for or history of a thromboembolic event must agree to receive prophylactic anticoagulation therapy (e.g., vitamin K) to keep INR in the range of 2-3
* No New York Heart Association class III-IV disease
* No blood donating during and for 1 week after completion of study therapy
* No uncontrolled infectious disease, autoimmune disease, or immunodeficiency
* No second malignancies within the past 3 years except surgically cured carcinoma in situ of the cervix, in situ breast cancer, incidental finding of stage T1a or T1b prostate cancer, and basal or squamous cell carcinoma of the skin
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* No Lapp lactase deficiency or history of glucose-galactose malabsorption

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No other prior intravenous chemotherapy for this cancer

  * For purposes of this protocol, the definition of intravenous chemotherapy also includes denileukin diftitox, antibodies, or antibody conjugates
* No prior splenectomy or splenic irradiation
* No concurrent topical corticosteroids

  * Concurrent systemic corticosteroids allowed for treatment of tumor flare reactions
* No radiation or drug-based therapy (including steroids) between registration and randomization
* No other concurrent drugs (including steroids) during the debulking regimen

  * Low-dose steroids as premedication allowed at the investigator's discretion
* No other concurrent anticancer treatments

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Overall survival
Progression-free survival as assessed by hematogenous disease criteria
Acute and late toxicity
Conversion rate
Rate of occurrence of second cancers at any site

CONTACTS AND LOCATIONS:
Overall Officials: Martine Bagot, MD, Study Chair — Hopital Saint-Louis
Locations (22):
- Austria (2):
  - Medical University of Graz, Graz
  - Medical University Vienna - General Hospital, Vienna
- Belgium (3):
  - Cliniques Universitaires St. Luc, Brussels
  - Hôpitaux Universitaires Bordet-Erasme - Institut Jules Bordet, Brussels
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
- Helsinky University Central Hospital - Skin & Allergy Hospital, Helsinki, Finland
- France (6):
  - Nouvel Hopital Estaing, Clermont-Ferrand, Cedex 1
  - Chu de Bordeaux - Hopital Du Haut Leveque, Bordeaux, Pessac Cedex
  - Chu Lyon - Centre Hospitalier Lyon Sud, Lyon, Pierre-Benite Cedex
  - Chu Amiens - Hopital Sud, Amiens
  - Hopital Saint-Louis, Paris
  - CHU de Reims - Hôpital Robert Debré, Reims
- Germany (3):
  - Charite - Universitaetsmedizin Berlin - Campus Mitte, Berlin
  - Johannes Gutenberg Universitaetskliniken, Mainz
  - Johannes Wesling Klinikum Minden, Minden
- Spain (2):
  - Csu de Bellvitge (Institut Catala D'Oncologia), L'Hospitalet de Llobregat
  - Hospital Universitario 12 De Octubre, Madrid
- UniversitaetsSpital Zurich - Division of Oncology, Zurich, Switzerland
- United Kingdom (4):
  - NHS Greater Glasgow and Clyde - Beatson West of Scotland Cancer Centre, Glasgow
  - Guy'S and St Thomas' Nhs - St Thomas Hospital, London
  - Christie Nhs Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust - City Hospital campus, Nottingham